CLINICAL TRIAL: NCT03629210
Title: Combination OZURDEX® & EyLea® vs. OZURDEX® Monotherapy in IncompLete-Responders wIth Diabetic Macular Edema (COLLIDE)
Brief Title: Combination OZURDEX® & EyLea® vs. OZURDEX® Monotherapy in IncompLete-Responders wIth Diabetic Macular Edema
Acronym: COLLIDE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study funding discontinued
Sponsor: Pradeepa Yoganathan (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor-Investigator, Pradeepa Yoganathan, Ophthalmologist, North Toronto Eye Care Laser and Eye Specialists
Organization: North Toronto Eye Care Laser and Eye Specialists (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLLIDE2018-05
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone; aflibercept

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 1:1 manner to one of the following groups:
  * Combination treatment (Group A): 50 participants will receive an intravitreal AFL (2.0 mg) injection and DEX implant (0.7 mg) injection within 0 to 8 days of each other.
  * Monotherapy treatment (Group B): 50 participants will receive DEX implant (0.7 mg) injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Treatment (Experimental): Combination treatment: Participants will receive intravitreal Eylea (AFL, 2.0 mg) injection and OZURDEX implant (0.7 mg) injection within 0 to 8 days of each other.
  Interventions: Drug: OZURDEX; Biological: Eylea
- Monotherapy (Active Comparator): Monotherapy treatment: Participants will receive OZURDEX implant (0.7 mg) injection.
  Interventions: Drug: OZURDEX

INTERVENTIONS:
Drug: OZURDEX — OZURDEX® (DEX implant, 0.7 mg) is a micro-ionized and non-preserved dexamethasone within a cylindrically-shaped 0.45 mm diameter x 6.5 mm length biodegradable Poly D, L-lactate-co-glycolic acid pellet allowing for sustained delivery dexamethasone into the vitreous cavity and retina following intravitreal injection. Health Canada has granted approval for use of DEX implant in the treatment of ME following central retinal vein occlusion, non-infectious uveitis affecting the posterior segment and pseudophakic DME in adult patients. (OZURDEX® Canadian Product Monograph, April 14, 2015). DEX implant will be provided as investigational treatment by Allergan Inc., Markham, ON, Canada.
  Other Names: DEX, dexamethasone
Biological: Eylea — EYLEA® (AFL 2.0 mg intravitreal injections) is an anti-VEGF treatment. AFL (2.0 mg) has received approval from Health Canada for the treatment of DME. Health Canada has also granted approval for AFL (2.0 mg) in the treatment of age-related macular degeneration, and ME secondary to retinal vein occlusion.
  Arms: Combination Treatment

SUMMARY:
COLLIDE is a multi-center, open-label, 1:1 randomized study looking at the effects of aflibercept (AFL; 2.0mg) plus OZURDEX (DEX; 0.7mg) implant combination therapy versus DEX monotherapy in phakic or pseudophakic eyes with center-involved DME that have demonstrated prior incomplete response to 3-6 anti-VEGF treatment in 3-9 months. The primary outcome will be 24 week central subfield thickness. Secondary outcomes include the change in ETDRS BCVA letters, number of re-injections and re-injection interval, proportion of eyes with 15- and 10- ETDRS letter gained/lost, proportion of eyes with PDR as per Optos color and FA at the study completion (24+/- 2 weeks) and OCT and OCT angiography biomarkers.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is a common cause of vision loss in patients with diabetes. The pathophysiology of DME is complex and likely multifactorial, where some of the most important features include the accumulation of advanced glycation end products, reactive oxygen species, protein kinase C and diacylglyceride activation, up-regulation of the renin-angiotensin-aldosterone system and up-regulation of vascular endothelial growth factor (VEGF). Additionally, inflammation has also been identified as an important etiological factor because breakdown of the retinal pigment epithelium - a physiologic barrier to fluid flow from the choriocapillaris and active retinal fluid pump, has been linked to increased levels of pro-inflammatory mediators including VEGF and processes that support leukostasis.

In Canada, LUCENTIS® (0.5 mg ranibizumab or RBZ, an anti-neovascular VEGF-A inhibitor, Novartis Pharmaceuticals Canada Inc.) was the first approved medical treatment for DME. Health Canada's decision for regulatory approval of RBZ (0.5 mg) for treatment of DME was based on 12-month results from the RESOLVE (Phase II trial investigating RBZ (0.3 mg or 0.5 mg) vs. sham injection) and RESTORE (Phase IIIb trial investigating RBZ (0.5 mg) + sham laser or RBZ (0.5 mg) + laser vs. laser + sham injection) trials. In the RESOLVE trial, pooled RBZ treatment arms resulted in significant and continuous improvement compared to sham treatment in both BCVA (mean improvement of 7.8 letters with RBZ treatment compared to a mean decline of 0.1 letters with sham treatment) and CRT (mean reduction of -194.2 µm with RBZ treatment vs. -48.4±153.4 µm with sham treatment). Similarly in the RESTORE trial, RBZ monotherapy and RBZ treatment with adjunctive laser yielded a statistically significantly greater mean average change in BCVA letter score compared to laser monotherapy through 12-months of study (+6.1 and +5.9 vs. +0.8 BCVA letters, respectively) along with a significantly greater improvement in CRT change from baseline vs. laser (-118.7 µm and -128.3 µm vs. -61.3 µm, respectively). Additionally, RBZ treatment arms in both RESOLVE and RESTORE demonstrated comparable safety with controls permitting conclusions that RBZ 0.5 mg is well-tolerated in the management of DME.

Diabetic Retinopathy Clinical Research Network (DRCR.net) published in 2015 their Protocol T: Comparison of RBZ with Eylea (Aflibercept or AFL, Regeneron Pharmaceuticals) and Avastin (Bevacizumab or BCZ, Roche) in DME. At 1 year, the patients treated with AFL had a statistically improved visual acuity of 13.3 letters as compared to BCZ (9.7 letters) and RBZ (11.2 letters). The same cohort of AFL treated DME had greater improvement on Ocular Coherence Tomography central subfield thickness with 169 micron change vs 101 um with BCZ and 147 um with RBZ. However, in all treatment arms, a large number of patients 46% required rescue laser therapy as per study protocol.

While anti-VEGF agents are a mainstay for the management of DME, a subgroup of eyes having partial or incomplete response to AVASTIN® (bevacizumab or BCZ), EYLEA® (intravitreal aflibercept injection or AFL) and RBZ exist.

RISE and RIDE, two phase III trials for registration of RBZ in the USA randomized DME patients on a basis of 1:1:1 to receive monthly 0.3 mg or 0.5 mg RBZ intravitreal treatments or sham injections over 24 months. Upon completion of the 24-month study (time point for primary efficacy outcome, namely the proportion of patients gaining ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters in BCVA from baseline), patients within the sham arm were eligible to receive delayed monthly 0.5 mg RBZ treatments over the next 12 months. Although strong vision gains were observed in patients originally randomized to RBZ arms at month 24 and sustained through month 36, sham controls receiving delayed RBZ treatment had vision improvements to a lesser extent than those receiving continuous RBZ treatment throughout the 36 month study, thereby suggesting benefits with initiation of DME treatment early in the course of DME management.

In a prospective study comparing the efficacy of monthly BCZ (1.5 mg) vs. monthly RBZ (0.5 mg) in eyes with baseline center-involved DME > 300 µm, Nepomuceno and colleagues reported 59% and 37% of eyes had persistent DME (> 275 µm) by week 48. Moreover, 28% and 14% of BCZ- and RBZ-treated eyes qualified for rescue therapy, respectively.

Results from the phase 3 VIVID and VISTA trials demonstrated that 42% eyes with central involved DME treated with Eylea (Aflibercept) 2.0 mg administered either every 4 or 8 weeks (after 5 initial monthly doses) failed to achieve 2-lines of vision gain.

In the RESOLVE and RESTORE trials there were 39.2% and 59.7% of RBZ-treated eyes that respectively failed to achieve 2-lines of vision gain at 12 months of study, while in RISE and RIDE, 23% of patients had CRT >250 µm and 40% of patients failed to achieve a best-corrected visual acuity (BCVA) ≥ 20/40 despite 2 years of monthly RBZ injections.

Adjunctive treatment regimens that offer ability to resolve DME and improve vision in eyes with incomplete response to anti-VEGF monotherapy will be of great value. Given that the treatment effects observed with delayed treatment in RISE and RIDE were less than that seen in the continuous (early) RBZ treatment arms, one may reason it is beneficial to readily identify eyes with incomplete response to anti-VEGF monotherapy to best allow functional vision improvement with an effective adjunctive treatment option.

Intravitreal corticosteroids may be useful in the treatment of DME because they block production of VEGF and other inflammatory mediators, inhibit leukostasis, and enhance the barrier function of vascular endothelial cell tight junctions. Off-label treatment with IVTA has been shown to be more effective than placebo in improving vision in patients with refractory DME. Sustained-release corticosteroids have been developed to reduce the need for frequent retreatments associated with anti-VEGF monotherapy regimens.

OZURDEX® (DEX implant; Allergan Inc. Irvine, CA, USA) is a sustained-release biodegradable implant approved for treatment of ME following central retinal vein occlusion, non-infectious uveitis affecting the posterior segment and pseudophakic DME in adult patients. DEX implant releases the corticosteroid dexamethasone, which possesses 5-6 times greater anti-inflammatory potency than triamcinolone, into the vitreous over a period of 6 months. In previous studies, DEX implant has demonstrated efficacy in the treatment of persistent DME, DME resistant to anti-VEGF treatment and DME in difficult-to-treat vitrectomized eyes. Recently, the results of two identical phase III, multi-center, international, masked, randomized, sham-controlled trials of DEX implants (0.35 mg and 0.7 mg) in DME demonstrated that an average of 4-5 DEX implant injections administered at ≥ 6-month intervals over 3 years provides rapid and sustained functional and anatomical improvements. Retreatment with the 0.7 mg DEX implant in phakic DME eyes was associated with significant 67.9% cataract-related adverse events and 59.2% cataract surgery rate vs. only 20.4% and 7.2% rates observed in sham-controls. These cataract-related adverse event rates are comparatively lower for a DEX implant than for other commonly used intravitreal corticosteroids. As such, a DEX implant may have a better benefit to risk safety profile. A meta-analysis on corticosteroid-induced IOP elevation for the three commonly used intravitreal corticosteroids including off-label KENALOG® (intravitreal triamcinolone acetonide or IVTA (4.0 mg), Bristol-Myers Squibb, Canada. Montreal, Quebec), DEX implant and RETISERT® (intravitreal fluocinolone acetonide or IFA (0.59 mg) non-biodegradable implant, Bausch & Lomb Canada Inc., Vaughan, Ontario) found the incidence of ocular hypertension to be lowest among eyes treated with DEX implant (15%) followed by IVTA (32%) and IFA (66%).

DRCR.net Protocol U studied the effect of adding Ozurdex to patients who had incomplete response to at least 3 anti-VEGF injections. The authors randomized 116 phakic and pseudophakic patients with DME to either Ozurdex plus RBZ or RBZ alone. Change in OCT subfoveal thickness was significantly different between both groups with 110 um reduction in the ozurdex arm vs 62 um in the monotherapy RBZ arm.

The present study seeks to compare the effects of a combination treatment regimen consisting of AFL (2.0 mg) + DEX implant vs. DEX implant monotherapy in phakic or pseudophakic eyes with center-involved DME deemed to have incomplete response to 3-6 prior anti-VEGF treatments.

It is hypothesized that phakic or pseudophakic center-involved DME eyes with incomplete response to 3-6 anti-VEGF injections (i.e., RBZ, BCZ or IAI) will show a greater reduction in central subfield thickness (CST) at 24 weeks when treated with a combination treatment regimen consisting of AFL (2.0 mg) and DEX implant (0.7 mg) vs. a monotherapy treatment regimen with DEX implant (0.7 mg).

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetic adult (≥18 years) patients
2. Known glycosylated haemoglobin (HbA1c) levels ≤ 11%
3. Screening Snellen Va / Baseline ETDRS BCVA between 20/20 - 20/320
4. Lens status: Phakic without significant cataract; <1+ nuclear sclerosis and <1+ posterior subcapsular or pseudophakic with intact posterior lens capsule and / or Nd:YAG laser capsulotomy that in the investigator's opinion is not likely to permit dislocation of DEX implant into the anterior chamber
5. Center-involved DME > 250 µm
6. Duration of DME ≤ 2 years
7. Eyes with intraocular pressure (IOP) ≤ 21 with or without treatment with < 2 topical IOP-lowering medications
8. Eyes with history of previous angle closure that have been successfully treated with either laser or surgical intervention are allowed as long as the visual fields and optic nerves have been stable for > 1 year prior to study entry
9. Demonstrated incomplete response to 3-6 prior intravitreal anti-VEGFs (AVASTIN®, LUCENTIS®, or EYLEA®; administered every 4 ± 2 weeks over 12-36 weeks (or 3-9 months)); incomplete response is defined herein as a treatment effect resulting in:

   1. < 25% reduction in central subfield thickness (CST) by SD-OCT during two recent visits OR
   2. < 10-letter (2 lines) increase in visual acuity compared to the baseline first anti-VEGF injection
10. If both eyes qualify, investigators can enrol the eye that has developed DME most recently.
11. Written informed patient consent

Exclusion Criteria:

1. Prior panretinal or macular laser treatments
2. Any Intravitreal injection prior to run-in phase
3. Previous vitrectomy
4. Any ocular condition that in the opinion of the investigator would not permit improvement of visual acuity with resolution of ME (e.g., epiretinal membrane, foveal atrophy, known macular ischemia, pigment abnormalities, dense subfoveal hard exudates and/or poor foveal architecture suggestive of photoreceptor loss)
5. Patients with retinal diseases, other than diabetes that can affect ME
6. HbA1c levels > 11%
7. Patient has suffered from a stroke in the last 3 months
8. Eyes with a history of advanced glaucoma (optic nerve head change consistent with glaucoma damage and / or glaucomatous visual field loss), uncontrolled ocular hypertension (baseline IOP > 21 mmHg despite use of ≥ 2 topical IOP-lowering medication)
9. Eyes with a history of steroid response (i.e., increase of ≥ 5 mmHg IOP following topical steroid treatment)
10. Patients with ACIOL (Anterior Chamber Intraocular Lens) or rupture of the posterior lens capsule that in the investigator's opinion is likely to permit dislocation of DEX implant into the anterior chamber
11. Female patients who are pregnant or breast feeding: all women of child bearing potential (i.e. women who are not surgically sterile or who have had one or more menstrual cycle in the previous 12 months) must have a negative pregnancy test prior to randomization, and must agree to use appropriate measures to avoid pregnancy during the trial period.
12. Patients who are unable to attend scheduled follow-up visits throughout the 24-week study
13. Use of systemic steroid, systemic anti-VEGF or pro-VEGF treatment within 4 months prior to enrolment or anticipated use during the study (these drugs are prohibited from use during the study)
14. Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
15. Patients with known hypersensitivity to any components of anti-VEGF or DEX implant
16. Patients using topical anti-inflammatory medication for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Central Subfield Thickness | At 24 Weeks
  Foveal central subfield (FCS) thickness is defined as the average thickness in the central 1mm diameter circle of the ETDRS grid.

SECONDARY OUTCOMES:
ETDRS BCVA letters | From Baseline to 24 Weeks
  Visual acuity measurement
Number of re-injections | At 24 Weeks
  Analyzing whether or not retreatment with the assigned intervention is required and how often in each group, comparatively
Proportion of eyes with 15- and 10-ETDRS letters gained/lost at study completion | 24 Weeks
  Visual Acuity
Proportion of study eyes with PDR as per Optos color and FA at the study completion | 24 Weeks
  Looking for proliferative diabetic retinopathy comparatively in each group
Ocular Coherence Tomography | 24 Weeks
  Medical imaging technique

CONTACTS AND LOCATIONS:
Overall Officials: Pradeepa Yoganathan, MD, FRCP(C), Principal Investigator — North Toronto Eye Care

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antcliff RJ, Marshall J. The pathogenesis of edema in diabetic maculopathy. Semin Ophthalmol. 1999 Dec;14(4):223-32. doi: 10.3109/08820539909069541. PMID 10758223
- [Background] Antonetti DA, Wolpert EB, DeMaio L, Harhaj NS, Scaduto RC Jr. Hydrocortisone decreases retinal endothelial cell water and solute flux coincident with increased content and decreased phosphorylation of occludin. J Neurochem. 2002 Feb;80(4):667-77. doi: 10.1046/j.0022-3042.2001.00740.x. PMID 11841574
- [Background] Boyer DS, Faber D, Gupta S, Patel SS, Tabandeh H, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex CHAMPLAIN Study Group. Dexamethasone intravitreal implant for treatment of diabetic macular edema in vitrectomized patients. Retina. 2011 May;31(5):915-23. doi: 10.1097/IAE.0b013e318206d18c. PMID 21487341
- [Background] Boyer DS, Yoon YH, Belfort R Jr, Bandello F, Maturi RK, Augustin AJ, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Three-year, randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1904-14. doi: 10.1016/j.ophtha.2014.04.024. Epub 2014 Jun 4. PMID 24907062
- [Background] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Background] Chang-Lin JE, Attar M, Acheampong AA, Robinson MR, Whitcup SM, Kuppermann BD, Welty D. Pharmacokinetics and pharmacodynamics of a sustained-release dexamethasone intravitreal implant. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):80-6. doi: 10.1167/iovs.10-5285. PMID 20702826
- [Background] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Funatsu H, Noma H, Mimura T, Eguchi S, Hori S. Association of vitreous inflammatory factors with diabetic macular edema. Ophthalmology. 2009 Jan;116(1):73-9. doi: 10.1016/j.ophtha.2008.09.037. PMID 19118698
- [Background] Gillies MC, Sutter FK, Simpson JM, Larsson J, Ali H, Zhu M. Intravitreal triamcinolone for refractory diabetic macular edema: two-year results of a double-masked, placebo-controlled, randomized clinical trial. Ophthalmology. 2006 Sep;113(9):1533-8. doi: 10.1016/j.ophtha.2006.02.065. Epub 2006 Jul 7. PMID 16828501
- [Background] Treatment techniques and clinical guidelines for photocoagulation of diabetic macular edema. Early Treatment Diabetic Retinopathy Study Report Number 2. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1987 Jul;94(7):761-74. doi: 10.1016/s0161-6420(87)33527-4. PMID 3658348
- [Background] Haller JA, Bandello F, Belfort R Jr, Blumenkranz MS, Gillies M, Heier J, Loewenstein A, Yoon YH, Jacques ML, Jiao J, Li XY, Whitcup SM; OZURDEX GENEVA Study Group. Randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with macular edema due to retinal vein occlusion. Ophthalmology. 2010 Jun;117(6):1134-1146.e3. doi: 10.1016/j.ophtha.2010.03.032. Epub 2010 Apr 24. PMID 20417567
- [Background] Hooper P, Boucher MC, Colleaux K, Cruess A, Greve M, Lam WC, Shortt S, Tourville E. Contemporary management of diabetic retinopathy in Canada: from guidelines to algorithm guidance. Ophthalmologica. 2014;231(1):2-15. doi: 10.1159/000354548. Epub 2013 Nov 12. PMID 24246998
- [Background] Kiddee W, Trope GE, Sheng L, Beltran-Agullo L, Smith M, Strungaru MH, Baath J, Buys YM. Intraocular pressure monitoring post intravitreal steroids: a systematic review. Surv Ophthalmol. 2013 Jul-Aug;58(4):291-310. doi: 10.1016/j.survophthal.2012.08.003. PMID 23768920
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Lazic R, Lukic M, Boras I, Draca N, Vlasic M, Gabric N, Tomic Z. Treatment of anti-vascular endothelial growth factor-resistant diabetic macular edema with dexamethasone intravitreal implant. Retina. 2014 Apr;34(4):719-24. doi: 10.1097/IAE.0b013e3182a48958. PMID 23975006
- [Background] Massin P, Bandello F, Garweg JG, Hansen LL, Harding SP, Larsen M, Mitchell P, Sharp D, Wolf-Schnurrbusch UE, Gekkieva M, Weichselberger A, Wolf S. Safety and efficacy of ranibizumab in diabetic macular edema (RESOLVE Study): a 12-month, randomized, controlled, double-masked, multicenter phase II study. Diabetes Care. 2010 Nov;33(11):2399-405. doi: 10.2337/dc10-0493. PMID 20980427
- [Background] Maturi RK, Glassman AR, Liu D, Beck RW, Bhavsar AR, Bressler NM, Jampol LM, Melia M, Punjabi OS, Salehi-Had H, Sun JK; Diabetic Retinopathy Clinical Research Network. Effect of Adding Dexamethasone to Continued Ranibizumab Treatment in Patients With Persistent Diabetic Macular Edema: A DRCR Network Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jan 1;136(1):29-38. doi: 10.1001/jamaophthalmol.2017.4914. PMID 29127949
- [Background] Medeiros MD, Alkabes M, Navarro R, Garcia-Arumi J, Mateo C, Corcostegui B. Dexamethasone intravitreal implant in vitrectomized versus nonvitrectomized eyes for treatment of patients with persistent diabetic macular edema. J Ocul Pharmacol Ther. 2014 Nov;30(9):709-16. doi: 10.1089/jop.2014.0010. Epub 2014 Sep 26. PMID 25259834
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Background] Miyamoto K, Khosrof S, Bursell SE, Rohan R, Murata T, Clermont AC, Aiello LP, Ogura Y, Adamis AP. Prevention of leukostasis and vascular leakage in streptozotocin-induced diabetic retinopathy via intercellular adhesion molecule-1 inhibition. Proc Natl Acad Sci U S A. 1999 Sep 14;96(19):10836-41. doi: 10.1073/pnas.96.19.10836. PMID 10485912
- [Background] Nepomuceno AB, Takaki E, Paes de Almeida FP, Peroni R, Cardillo JA, Siqueira RC, Scott IU, Messias A, Jorge R. A prospective randomized trial of intravitreal bevacizumab versus ranibizumab for the management of diabetic macular edema. Am J Ophthalmol. 2013 Sep;156(3):502-510.e2. doi: 10.1016/j.ajo.2013.04.026. Epub 2013 Jun 21. PMID 23795985
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Pacella E, Vestri AR, Muscella R, Carbotti MR, Castellucci M, Coi L, Turchetti P, Pacella F. Preliminary results of an intravitreal dexamethasone implant (Ozurdex(R)) in patients with persistent diabetic macular edema. Clin Ophthalmol. 2013;7:1423-8. doi: 10.2147/OPTH.S48364. Epub 2013 Jul 16. PMID 23901252
- [Background] Maturi RK. (2013). Combined steroids, anti-VEGFs show promise in DME. Ophthalmology Times.
- [Background] Maturi RK. (2014). Ozurdex as adjunct to avastin compared to avastin alone in treatment of patients with diabetic macular edema. ClinicalTrials.gov Identifier: NCT01309451 (http://clinicaltrials.gov/ct2/show/record/NCT01309451)
- [Background] Tamura H, Miyamoto K, Kiryu J, Miyahara S, Katsuta H, Hirose F, Musashi K, Yoshimura N. Intravitreal injection of corticosteroid attenuates leukostasis and vascular leakage in experimental diabetic retina. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1440-4. doi: 10.1167/iovs.04-0905. PMID 15790913
- [Background] Wang K, Wang Y, Gao L, Li X, Li M, Guo J. Dexamethasone inhibits leukocyte accumulation and vascular permeability in retina of streptozotocin-induced diabetic rats via reducing vascular endothelial growth factor and intercellular adhesion molecule-1 expression. Biol Pharm Bull. 2008 Aug;31(8):1541-6. doi: 10.1248/bpb.31.1541. PMID 18670086
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915